CLINICAL TRIAL: NCT05912829
Title: Evaluation of Two Different Intraocular Lens Models After Lens Implantation Using the Yamane Technique
Brief Title: Comparison of Two Different Intraocular Lenses Implanted With Yamane Technique
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Kepler University of Linz (Other)
Responsible Party: Sponsor
Other Study IDs: KUK-Ophthalmology-012
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Secondary Cataract Surgery; Aphakia; Complicated Cataract Surgery
MeSH Terms: conditions — Aphakia | interventions — Microscopy, Acoustic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Kowa Group: Patients who had a Kowa lens implanted using the Yamane technique
  Interventions: Device: IOL Master 700; Device: Casia-2; Device: MS-39; Device: OSIRIS; Device: Autorefractor; Diagnostic Test: Subjective Refraction; Diagnostic Test: Biomicroscopy
- Johnson: Patients who had the ZA9003 (J&J) lens implanted using the Yamane technique
  Interventions: Device: IOL Master 700; Device: Casia-2; Device: MS-39; Device: OSIRIS; Device: Autorefractor; Diagnostic Test: Subjective Refraction; Diagnostic Test: Biomicroscopy

INTERVENTIONS:
Device: IOL Master 700 — Biometry using the IOL Master 700
Device: Casia-2 — Anterior segment-OCT to evaluate lens tilt
Device: MS-39 — Corneal Topography using the MS-39
Device: OSIRIS — Abberometry using the OSIRIS-Abberometer
Device: Autorefractor — Evaluation of Refraction using an Autorefractor
Diagnostic Test: Subjective Refraction — Refraction performed by experienced staff
Diagnostic Test: Biomicroscopy — Slit Lamp Examination

SUMMARY:
In case of instability or rupture of capsular bag occurs during cataract surgery, Yamane technique is one of the options to fix intracocularlens' haptics. Yamane technique uses a double-needle technique that seamlessly fixes the haptics intrascleral by creating a scleral tunnel.

Aberrations, IOL tilting or even dislocations might occur and influence the final outcome of IOL implantation.

The aim of this study is the evaluation of the postoperative tilt of Kowa PU6AS using Yamane technique. Furthermore of the corrected and uncorrected visual acuity and the anterior chamber depth are being developed.

DETAILED DESCRIPTION:
During uncomplicated cataract surgery, an intraocular lens (IOL) is implanted into the patient's capsular bag. If increased instability or rupture of this capsular bag occurs due to aggravated intraoperative conditions or IOL dislocation, several options are available to the surgeon to correct the aphakia, all characterized by their respective advantages and disadvantages, but with no clear superiority of any one method.

The popular Yamane technique, or "flanged IOL fixation", uses a double-needle technique that seamlessly fixes the haptics intrascleral by creating a scleral tunnel using two 30-gauge needles.

Examples of lenses used for this purpose are the TECNIS ZA9003 (Johnson&Johnson, USA) and the Kowa PU6AS (Kowa, Japan). Another approach is the Carlevale FIL-SSF IOL (Soleko, Italy), which was developed specifically for use in aphakia with lack of capsular stability.

All types of implantation are not immune to aberrations, tilting or even dislocation. Many factors influence the final outcome of IOL implantation, be it the optimal choice of intraocular lens power, the surgeon's experience regarding fixation in more challenging eyes, or individual anatomical conditions. As part of quality assurance, an evaluation of monthly and six-monthly data will now be performed. The aim of this study is the evaluation of the postoperative tilt of the Kowa PU6AS in Yamane technique, as well as the evaluation of the corrected and uncorrected visual acuity and the anterior chamber depth within the clinical quality management.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age: 21 Years
* planned or performed lens implantation using the Kowa PU6AS or the Johnson & Johnson ZA9003 using the Yamane technique
* signed patient consent form

Exclusion Criteria:

* best corrected visual acuity >0.1 (Snellen)
* pregnancy

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Only patients who are undergoing (underwent)routine secondary cataract surgery will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Tilt | 6 Weeks
  Postoperative Tilt
Autorefraction | 6 Weeks
  Refraction using an automated refractor
Subjective Refraction | 6 Weeks
  Refraction performed by experienced staff
Best corrected visual acuity | 6 Weeks
  Measurement performed by experienced staff
uncorrected visual acuity | 6 Weeks
  Measurement performed by experienced staff

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Bolz, MD, Study Chair — JKU Linz
Locations (2):
- Austria (2):
  - Department for Ophthalmology and Optometry, Kepler University Hospital GmbH, Johannes Kepler University Linz, Linz, Upper Austria
  - Department for Ophthalmology and Optometry, Linz, Upper Austria

IPD SHARING:
Plan to Share IPD: No